CLINICAL TRIAL: NCT02265224
Title: Comparative Bioavailability Study of N-acetyl-cysteine (NAC) 600 mg Uncoated Tablets vs. NAC 600 mg Film-coated Tablets in Healthy Male and Female Volunteers
Brief Title: Bioequivalence Study of Two Different Formulations of N-acetyl-cysteine (NAC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zambon SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Z7169J02; CRO-PK-14-286 (Other: Cross Research SA)
Record Dates: First submitted 2014-10-03; First posted 2014-10-15 (Estimated); Results first posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: no Condition
Keywords: healthy volunteers
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Test - Reference (Experimental): N-acetylcysteine (NAC) 600 mg uncoated tablet (single dose) followed by NAC 600 mg film-coated tablet (single dose)
  Interventions: Drug: N-acetylcysteine
- Reference - Test (Active Comparator): N-acetylcysteine (NAC) 600 mg film-coated tablet (single dose) followed by NAC 600 mg uncoated tablet (single dose)
  Interventions: Drug: N-acetylcysteine

INTERVENTIONS:
Drug: N-acetylcysteine — The product was administered according to the randomisation list and cross-over design, with 150 mL of still mineral water under fasting conditions on study day 1 of periods 1 or 2 at 8:00±1 h.
  Other Names: Fluimucil uncoated tablets

SUMMARY:
Study primary Objective:

- To evaluate the bioequivalent rate (Cmax) and extent (AUC0-t) of absorption of N-acetyl-cysteine 600 mg uncoated tablets vs. N-acetyl-cysteine 600 mg film-coated tablets (NAC) in healthy male and female volunteers.

Study secondary objectives:

* To describe the pharmacokinetic (PK) profile of NAC in plasma after single dose administration of NAC 600 mg uncoated tablets vs. NAC 600 mg film-coated tablets;
* to collect safety and tolerability data after single dose administration of NAC 600 mg uncoated tablets vs. NAC 600 mg film-coated tablets.

DETAILED DESCRIPTION:
This is single centre, single dose, open, randomised, cross-over, two-stage bioequivalence study to compare two different oral formulations of NAC.

The study has been conducted in healthy volunteers of both genders, in one single dose of both formulations.

The initial 48 subjects were sufficient to satisfy the study objectives on the basis of the ad interim preliminary bioequivalence test. The study was then considered as concluded and the second stage did not take place.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent: signed written informed consent before inclusion in the study
2. Sex and age: males and females,18-55 years old, inclusive
3. Body Mass Index (BMI): 18.5-30 kg/m2, inclusive
4. Vital signs: systolic blood pressure (SBP) 100-139 mmHg, diastolic blood pressure (DBP) 50-89 mmHg, heart rate (HR) 50-90 bpm, measured after 5 min of rest in the sitting position
5. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the entire study
6. Contraception and fertility (females only): females of child-bearing potential and with an active sexual life must be using at least one of the following reliable methods of contraception:

   * Hormonal oral, implantable, transdermal, or injectable contraceptives for at least 2 months before the screening visit
   * A non-hormonal intrauterine device or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide for at least 2 months before the screening visit
   * A male sexual partner who agrees to use a male condom with spermicide
   * A sterile sexual partner Female participants of non-child-bearing potential or in post-menopausal status for at least 1 year will be admitted.

For all female subjects, pregnancy test result must be negative at screening (serum β-HCG test) and day -1 (urine test).

Exclusion Criteria:

1. Electrocardiogram (ECG 12-leads, supine position): clinically significant abnormalities
2. Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the study
3. Laboratory analyses: clinically significant abnormal laboratory values indicative of physical illness
4. Allergy: ascertained or presumptive hypersensitivity to the active principle and/or formulations' ingredients; history of anaphylaxis to drugs or allergic reactions in general, which the investigator considers may affect the outcome of the study
5. Diseases: significant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine or neurological diseases that may interfere with the aim of the study
6. Medications: medications, including over the counter (OTC) medications and herbal remedies for 2 weeks before the start of the study. Hormonal contraceptives for females will be allowed
7. Investigative drug studies: participation in the evaluation of any investigational product for 3 months before this study. The 3-month interval is calculated as the time between the first calendar day of the month that follows the last visit of the previous study and the first day of the present study
8. Blood donation: blood donations for 3 months before this study
9. Drug, alcohol, caffeine, tobacco: history of drug, alcohol [>1 drink/day for females and >2 drinks/day for males, defined according to the USDA Dietary Guidelines 2010], caffeine (>5 cups coffee/tea/day) or tobacco abuse (≥6 cigarettes/day)
10. Drug test: positive result at the drug test at screening or day-1
11. Alcohol test: positive alcohol breath test at day -1
12. Diet: abnormal diets (<1600 or >3500 kcal/day) or substantial changes in eating habits in the 4 weeks before this study; vegetarians
13. Pregnancy (females only): positive or missing pregnancy test at screening or day -1, pregnant or lactating women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milko Radicioni, MD, Principal Investigator — Cross Research SA

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 48 healthy subjects were included in the study, as planned, and received test and reference treatment according to the cross-over design.
Pre-assignment Details: Subjects were assigned to a sequence of treatments (TR or RT) according to the randomisation list. Randomisation number was given to the subjects on study day -1, Period 1, and was used to assign the treatment sequence according to the randomisation list.
  The randomisation list was computer-generated by the Contract Research Organisation (CRO) Biometry Unit, using the PLAN procedure of SAS® version 9.3 (TS1M1) (24). The randomisation list was supplied to the Phase I Unit before study start.
Groups:
- Enrolled Subjects Set: According to the crossover design, all the enrolled subjects received both NAC formulations based on the randomization schedule.Two single doses of 600 mg of NAC (one with test and one with reference formulation) were administered to each volunteer in two subsequent study periods (morning of day 1), separated by a wash-out interval of at least 5 days.
Period: Overall Study
Arm/Group | Enrolled Subjects Set
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Enrolled set: All subjects included in the interventional phase of the study. The enrolment was performed through randomised allocation to a treatment sequence.
Groups:
- Enrolled Subjects Set: According to the crossover design, all the enrolled subjects received both NAC formulations based on the randomization schedule. Two single doses of 600 mg of NAC (one with test and one with reference formulation) were administered to each volunteer in two subsequent study periods (morning of day 1), separated by a wash-out interval of at least 5 days.
Arm/Group | Enrolled Subjects Set
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 48
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 47
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Switzerland | 48

OUTCOME MEASURES:

1. Primary Outcome: Cmax of NAC After Single Dose Administration of Test and Reference
Description: Cmax is the maximum concentration level of the drug reached in plasma.
Time Frame: 0-24h (5,15, 30, 45, 60, 75, 90 min and 2, 3, 4, 6, 8, 12, 16 and 24 h postdose)
Population: PK set: all randomised subjects who fulfilled the study protocol requirements in terms of investigational medicinal product intake and had evaluable PK data readouts for the planned treatment comparisons, with no major deviations that could affect the PK results.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Test: N-acetylcysteine (NAC) 600 mg uncoated tablet (single dose). The product was administered according to the randomisation list and cross-over design, with 150 mL of still mineral water under fasting conditions on study day 1 of periods 1 or 2 at 8:00±1 h.
- Reference: N-acetylcysteine (NAC) 600 mg film-coated tablet (single dose). The product was administered according to the randomisation list and cross-over design, with 150 mL of still mineral water under fasting conditions on study day 1 of periods 1 or 2 at 8:00±1 h.
Arm/Group | Test | Reference
Number analyzed (Participants) | 48 | 48
ng/mL | 2804.38 (899.47) | 3215.63 (1382.02)
Statistical Analysis 1: Comparison: Test vs Reference; Test type: Equivalence — The statistical analysis took into account treatment, period, sequence and subject (sequence) as sources of variation. Acceptance criterion for bioequivalence was that the 94.12% confidence interval for the ratio between test and reference of the geometric means of the parameters under consideration fell within the 80.00-125.00% range, according to the current guidelines for bioequivalence studies and to the Pocock α spending function; p = 0.0136, ANOVA — p value for treatment effect; Geometric means ratio = 89.81, 94.12% CI 2-sided [82.82 to 97.40]

2. Primary Outcome: AUC0-t of NAC After Single Dose Administration of Test and Reference
Description: AUC0-t is the Area under the concentration-time curve from time zero to time t, calculated with the linear trapezoidal summation from time 0 to the last measurable data point.
Time Frame: 0-24h (5,15, 30, 45, 60, 75, 90 min and 2, 3, 4, 6, 8, 12, 16 and 24 h postdose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL*h
Arm/Group | Test | Reference
Number analyzed (Participants) | 48 | 48
ng/mL*h | 10637.87 (3100.94) | 11773.11 (3775.43)
Statistical Analysis 1: Comparison: Test vs Reference; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0047, ANOVA; p value for treatment effect; Geometric means ratio = 90.79, 94.12% CI 2-sided [85.25 to 96.69]

3. Secondary Outcome: AUC0-∞ of NAC After Single Dose Administration of Test and Reference
Description: AUC0-∞ is the area under the concentration-time curve extrapolated to infinity, calculated, if feasible, as AUC0-t + Ct/λz, where Ct is the last measurable drug concentration.
Time Frame: 0-24h (5,15, 30, 45, 60, 75, 90 min and 2, 3, 4, 6, 8, 12, 16 and 24 h postdose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL*h
Arm/Group | Test | Reference
Number analyzed (Participants) | 48 | 48
ng/mL*h | 12586.17 (3577.24) | 13739.43 (4190.59)
Statistical Analysis 1: Comparison: Test vs Reference; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0095, ANOVA — p value for treatment effect; Geometric means ratio = 91.86, 94.12% CI 2-sided [86.45 to 97.61]

4. Secondary Outcome: Tmax of NAC After Single Dose Administration of Test and Reference
Description: time to achieve the maximum concentration level of the drug in plasma.
Time Frame: 0-24h (5,15, 30, 45, 60, 75, 90 min and 2, 3, 4, 6, 8, 12, 16 and 24 h postdose)
Measure: Median (Full Range); unit: hours
Arm/Group | Test | Reference
Number analyzed (Participants) | 48 | 48
hours | 1.00 [0.50 to 3.00] | 1.00 [0.25 to 3.00]
Statistical Analysis 1: Comparison: Test vs Reference; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.5050, Friedman test

5. Secondary Outcome: t1/2 of NAC After Single Dose Administration of Test and Reference
Description: Half-life (t1/2) is the time to halve the plasma concentration level of the drug.
Time Frame: 0-24h (5,15, 30, 45, 60, 75, 90 min and 2, 3, 4, 6, 8, 12, 16 and 24 h postdose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Test | Reference
Number analyzed (Participants) | 48 | 48
hours | 14.11 (4.16) | 13.59 (2.69)

6. Secondary Outcome: Lambda Zeta of NAC After Single Dose Administration of Test and Reference
Description: Lambda zeta is the terminal elimination rate constant. Individual estimate of the terminal elimination rate constant can be calculated using log-linear regression of the terminal portions of the plasma concentration-versus-time curves.
Time Frame: 0-24h (5,15, 30, 45, 60, 75, 90 min and 2, 3, 4, 6, 8, 12, 16 and 24 h postdose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Test | Reference
Number analyzed (Participants) | 48 | 48
1/h | 0.05 (0.01) | 0.05 (0.01)

7. Secondary Outcome: Frel of NAC After Single Dose Administration of Test and Reference
Description: Frel is the relative bioavailability, calculated as ratio AUC0-t (test)/ AUC0-t (reference)
Time Frame: 0-24h (5,15, 30, 45, 60, 75, 90 min and 2, 3, 4, 6, 8, 12, 16 and 24 h postdose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage
Groups:
- Enrolled Subjects Set: According to the crossover design, all the enrolled subjects received both NAC formulations based on the randomization schedule.
Arm/Group | Enrolled Subjects Set
Number analyzed (Participants) | 48
percentage | 92.82 (18.05)

ADVERSE EVENTS:
Time Frame: From the beginning of screening days ( day -21 ) up to Final Visit (Day 2).
Arm/Group | Test - Reference | Reference - Test
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 4/48 | 2/48
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test - Reference (N=48) | Reference - Test (N=48)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations and Caveats not specified

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No